CLINICAL TRIAL: NCT01430663
Title: Diagnosing Pulmonary Aspergillosis in Patients With Hematological Malignancies: A Multicentre Prospective Evaluation of an Aspergillus PCR Assay and a Galactomannan ELISA in Bronchoalveolar Lavage Samples
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dieter Buchheidt, Prof. Dr. med., Heidelberg University
Other Study IDs: AGIHO BAL GM PCR 2007
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Invasive Aspergillosis
Keywords: aspergillosis; bronchoalveolar lavage; galactomannan; pcr; hematological patients
MeSH Terms: conditions — Aspergillosis; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hematological patients with proven or probable aspergillosis
- Hematological patients with possible aspergillosis

SUMMARY:
Diagnosing invasive pulmonary aspergillosis (IPA) remains a challenge in patients (pts) with hematological malignancies. The clinical significance of testing bronchoalveolar lavage (BAL) samples both with polymerase chain reaction (PCR) and Aspergillus galactomannan (GM) ELISA is unclear, and the BAL cutoff for GM has not been clearly defined yet. Using a validated nested PCR assay and a GM ELISA, we prospectively examine BAL samples from hematological patients at high risk of PA.

ELIGIBILITY:
Inclusion Criteria:

- hematological patients with lung infiltrates at high risk for invasive aspergillosis

Exclusion Criteria:

- patients without informed consent

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hematological patients at high risk for invasive aspergillosis
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2007-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Clinical significance of biomarker based diagnostic investigation in suspected invasive aspergillosis | up to 18 months

SECONDARY OUTCOMES:
Evaluation of diagnostic and therapeutic intervention concerning antifungal treatment with regard to outcome (overall survival, in months) of a fungal infection | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Buchheidt, MD, Principal Investigator — Mannheim University Hospital
Locations (9):
- Innsbruck University Hospital, Innsbruck, Austria
- Germany (8):
  - Cologne University Hospital, Cologne
  - Erlangen University Hospital, Erlangen
  - General Hospital Frankfurt (Oder), Frankfurt (Oder)
  - Freiburg University Hospital, Freiburg im Breisgau
  - Halle University Hospital, Halle
  - Herne University Hospital, Herne
  - Mannheim University Hospital, Mannheim
  - Würzburg University Hospital, Würzburg

REFERENCES:
- [Background] Skladny H, Buchheidt D, Baust C, Krieg-Schneider F, Seifarth W, Leib-Mosch C, Hehlmann R. Specific detection of Aspergillus species in blood and bronchoalveolar lavage samples of immunocompromised patients by two-step PCR. J Clin Microbiol. 1999 Dec;37(12):3865-71. doi: 10.1128/JCM.37.12.3865-3871.1999. PMID 10565898
- [Background] Buchheidt D, Baust C, Skladny H, Ritter J, Suedhoff T, Baldus M, Seifarth W, Leib-Moesch C, Hehlmann R. Detection of Aspergillus species in blood and bronchoalveolar lavage samples from immunocompromised patients by means of 2-step polymerase chain reaction: clinical results. Clin Infect Dis. 2001 Aug 15;33(4):428-35. doi: 10.1086/321887. Epub 2001 Jul 6. PMID 11462176
- [Background] Spiess B, Buchheidt D, Baust C, Skladny H, Seifarth W, Zeilfelder U, Leib-Mosch C, Morz H, Hehlmann R. Development of a LightCycler PCR assay for detection and quantification of Aspergillus fumigatus DNA in clinical samples from neutropenic patients. J Clin Microbiol. 2003 May;41(5):1811-8. doi: 10.1128/JCM.41.5.1811-1818.2003. PMID 12734210
- [Background] Hummel M, Spiess B, Cornely OA, Dittmer M, Morz H, Buchheidt D. Aspergillus PCR testing: results from a prospective PCR study within the AmBiLoad trial. Eur J Haematol. 2010 Aug;85(2):164-9. doi: 10.1111/j.1600-0609.2010.01452.x. Epub 2010 Apr 1. PMID 20374275